CLINICAL TRIAL: NCT00992927
Title: Comparative Study for the Efficacy of Capsule-Preserving Versus Capsule-Rupturing Intra-articular Hydraulic Distension in Patients With Painful Stiff Shoulders
Brief Title: Should the Joint Capsule of the Painful Stiff Shoulder be Ruptured During Intra-articular Hydraulic Distension?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sun Gun Chung/Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUH-RM-SGChung-IHD-01
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Adhesive Capsulitis
Keywords: Injections, Intra-Articular; Range of Motion, Articular; Pain
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPIHD (Experimental): Capsule-Preserving Intra-articular Hydraulic Distension (CPIHD) infuses as much volume as possible during the distension without rupturing the capsule.
  Interventions: Procedure: Capsule-Preserving Intra-articular Hydraulic Distension
- CRIHD (Active Comparator): Capsule-Rupturing Intra-articular Hydraulic Distension (CRIHD) infuses fluid into the joint space until the rupture of the capsule is observed.
  Interventions: Procedure: Capsule-Rupturing Intra-articular Hydraulic Distension

INTERVENTIONS:
Procedure: Capsule-Preserving Intra-articular Hydraulic Distension — Capsule-Preserving Intra-articular Hydraulic Distension (CPIHD) infuses as much volume as possible during the distension without rupturing the capsule.
  Arms: CPIHD
Procedure: Capsule-Rupturing Intra-articular Hydraulic Distension — Capsule-Rupturing Intra-articular Hydraulic Distension (CRIHD) infuses fluid into the joint space until the rupture of the capsule is observed.
  Arms: CRIHD

SUMMARY:
The purpose of the study is to compare the efficacy of intra-articular hydraulic distension (IHD) for the treatment of painful stiff shoulders between capsule-rupturing and capsule-preserving IHDs.

DETAILED DESCRIPTION:
The Painful stiff shoulder (PSS), or the adhesive capsulitis, involves stiff and contracted joint capsule from fibrosis in the glenohumeral joint. Intra-articular hydraulic distension (IHD) enlarges the stiffened capsule by deforming it with excessive volume and pressure within the joint space. Although IHD is one of the most common treatment options for the PSS, the diversity of the IHD technique spans wide range. Specifically, it is not generally agreed as for which, between capsule-rupturing and capsule-preserving IHDs, is superior for PSS treatment. Capsule-preserving IHD might fail to infuse sufficient amount of fluid to avoid rupture, thus producing less satisfactory outcomes. However, we devised in our previous study a novel technique that enabled a physician to infuse the possible largest volume without rupturing the capsule. By employing the technique, we aim to compare the clinical efficacy of capsule-rupturing versus capsule-preserving IHDs in patients with PSSs.

ELIGIBILITY:
Inclusion Criteria:

* shoulder discomfort for at least one month
* limited range of motion of the glenohumeral joint in at least two directions

Exclusion Criteria:

* systemic inflammatory joint disease
* radiological evidence of bony abnormality of the shoulder
* full-thickness rotator cuff tear
* acute systemic medical illness
* history of major trauma or surgery involving the shoulder
* contraindication to intra-articular, local anesthestic injection

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Gun Chung, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Buchbinder R, Green S, Forbes A, Hall S, Lawler G. Arthrographic joint distension with saline and steroid improves function and reduces pain in patients with painful stiff shoulder: results of a randomised, double blind, placebo controlled trial. Ann Rheum Dis. 2004 Mar;63(3):302-9. doi: 10.1136/ard.2002.004655. PMID 14962967
- [Background] Uhthoff HK, Boileau P. Primary frozen shoulder: global capsular stiffness versus localized contracture. Clin Orthop Relat Res. 2007 Mar;456:79-84. doi: 10.1097/BLO.0b013e318030846d. PMID 17179778
- [Background] Noel E, Thomas T, Schaeverbeke T, Thomas P, Bonjean M, Revel M. Frozen shoulder. Joint Bone Spine. 2000;67(5):393-400. PMID 11143905
- [Background] Hannafin JA, Chiaia TA. Adhesive capsulitis. A treatment approach. Clin Orthop Relat Res. 2000 Mar;(372):95-109. PMID 10738419
- [Background] Rodeo SA, Hannafin JA, Tom J, Warren RF, Wickiewicz TL. Immunolocalization of cytokines and their receptors in adhesive capsulitis of the shoulder. J Orthop Res. 1997 May;15(3):427-36. doi: 10.1002/jor.1100150316. PMID 9246090
- [Background] Hand GC, Athanasou NA, Matthews T, Carr AJ. The pathology of frozen shoulder. J Bone Joint Surg Br. 2007 Jul;89(7):928-32. doi: 10.1302/0301-620X.89B7.19097. PMID 17673588
- [Background] Amoretti N, Grimaud A, Brocq O, Roux C, Dausse F, Fournol M, Chevallier P, Bruneton JN. Shoulder distension arthrography in adhesive capsulitis. Clin Imaging. 2006 Jul-Aug;30(4):254-6. doi: 10.1016/j.clinimag.2006.01.022. PMID 16814141
- [Background] Gavant ML, Rizk TE, Gold RE, Flick PA. Distention arthrography in the treatment of adhesive capsulitis of the shoulder. J Vasc Interv Radiol. 1994 Mar-Apr;5(2):305-8. doi: 10.1016/s1051-0443(94)71488-3. PMID 8186599
- [Background] Ibrahim T, Rahbi H, Beiri A, Jeyapalan K, Taylor GJ. Adhesive capsulitis of the shoulder: the rate of manipulation following distension arthrogram. Rheumatol Int. 2006 Nov;27(1):7-9. doi: 10.1007/s00296-006-0160-1. Epub 2006 Jul 27. PMID 16871412
- [Background] Rizk TE, Gavant ML, Pinals RS. Treatment of adhesive capsulitis (frozen shoulder) with arthrographic capsular distension and rupture. Arch Phys Med Rehabil. 1994 Jul;75(7):803-7. PMID 8024429
- [Background] ANDREN L, LUNDBERG BJ. TREATMENT OF RIGID SHOULDERS BY JOINT DISTENSION DURING ARTHROGRAPHY. Acta Orthop Scand. 1965;36:45-53. doi: 10.3109/17453676508989370. No abstract available. PMID 14308098
- [Background] Ekelund AL, Rydell N. Combination treatment for adhesive capsulitis of the shoulder. Clin Orthop Relat Res. 1992 Sep;(282):105-9. PMID 1516300
- [Background] Mulcahy KA, Baxter AD, Oni OO, Finlay D. The value of shoulder distension arthrography with intraarticular injection of steroid and local anaesthetic: a follow-up study. Br J Radiol. 1994 Mar;67(795):263-6. doi: 10.1259/0007-1285-67-795-263. PMID 8130999
- [Background] Vad VB, Sakalkale D, Warren RF. The role of capsular distention in adhesive capsulitis. Arch Phys Med Rehabil. 2003 Sep;84(9):1290-2. doi: 10.1016/s0003-9993(03)00261-2. PMID 13680563
- [Background] Lee KJ, Lee HD, Chung SG. Real-time pressure monitoring of intraarticular hydraulic distension for painful stiff shoulders. J Orthop Res. 2008 Jul;26(7):965-70. doi: 10.1002/jor.20535. PMID 18271012
- [Background] Carette S, Moffet H, Tardif J, Bessette L, Morin F, Fremont P, Bykerk V, Thorne C, Bell M, Bensen W, Blanchette C. Intraarticular corticosteroids, supervised physiotherapy, or a combination of the two in the treatment of adhesive capsulitis of the shoulder: a placebo-controlled trial. Arthritis Rheum. 2003 Mar;48(3):829-38. doi: 10.1002/art.10954. PMID 12632439
- [Background] Jacobs LG, Barton MA, Wallace WA, Ferrousis J, Dunn NA, Bossingham DH. Intra-articular distension and steroids in the management of capsulitis of the shoulder. BMJ. 1991 Jun 22;302(6791):1498-501. doi: 10.1136/bmj.302.6791.1498. PMID 1855018
- [Background] Piotte F, Gravel D, Moffet H, Fliszar E, Roy A, Nadeau S, Bedard D, Roy G. Effects of repeated distension arthrographies combined with a home exercise program among adults with idiopathic adhesive capsulitis of the shoulder. Am J Phys Med Rehabil. 2004 Jul;83(7):537-46; quiz 547-9. doi: 10.1097/01.phm.0000130030.73449.60. PMID 15213478
- [Background] Lundberg BJ. The frozen shoulder. Clinical and radiographical observations. The effect of manipulation under general anesthesia. Structure and glycosaminoglycan content of the joint capsule. Local bone metabolism. Acta Orthop Scand Suppl. 1969;119:1-59. No abstract available. PMID 4952729
- [Background] Neer CS 2nd, Satterlee CC, Dalsey RM, Flatow EL. The anatomy and potential effects of contracture of the coracohumeral ligament. Clin Orthop Relat Res. 1992 Jul;(280):182-5. PMID 1611740
- [Background] Omari A, Bunker TD. Open surgical release for frozen shoulder: surgical findings and results of the release. J Shoulder Elbow Surg. 2001 Jul-Aug;10(4):353-7. doi: 10.1067/mse.2001.115986. PMID 11517365
- [Background] Ozaki J, Nakagawa Y, Sakurai G, Tamai S. Recalcitrant chronic adhesive capsulitis of the shoulder. Role of contracture of the coracohumeral ligament and rotator interval in pathogenesis and treatment. J Bone Joint Surg Am. 1989 Dec;71(10):1511-5. PMID 2592391
- [Background] Uitvlugt G, Detrisac DA, Johnson LL, Austin MD, Johnson C. Arthroscopic observations before and after manipulation of frozen shoulder. Arthroscopy. 1993;9(2):181-5. doi: 10.1016/s0749-8063(05)80371-8. PMID 8461078
- [Background] Warner JJ, Allen A, Marks PH, Wong P. Arthroscopic release for chronic, refractory adhesive capsulitis of the shoulder. J Bone Joint Surg Am. 1996 Dec;78(12):1808-16. doi: 10.2106/00004623-199612000-00003. PMID 8986657
- [Background] Wiley AM. Arthroscopic appearance of frozen shoulder. Arthroscopy. 1991;7(2):138-43. doi: 10.1016/0749-8063(91)90098-i. PMID 2069623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Dates: from Mar 2008 until Oct 2009 Type of Location: outpatient clinic at a university hospital Method of Recruitment: informed consent from eligible patients
Pre-assignment Details: Participants with other diagnoses than the painful stiff shoulder, such as full-thickness rotator cuff tear, osteoarthritis and others, were excluded from the trial when the final diagnosis was determined.
Period: Overall Study
Arm/Group | CPIHD | CRIHD
Started | 32 | 22
Completed | 32 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPIHD | CRIHD | Total
Number analyzed (Participants) | 32 | 22 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 11 | 4 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 61.09 (10.621) | 56.55 (9.521) | 59.24 (10.343)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 11 | 6 | 17
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 32 | 22 | 54
Pain Measured by Visual Analogue Scale (VAS) [Mean (Standard Deviation); unit: cm] — 1. before intervention for all participants
  2. using 10cm horizontal visual analog scale
  3. best: 0cm (no pain)
  4. worst: 10cm (worst pain)
  cm | 6.87 (3.01) | 7.17 (2.09) | 6.99 (2.65)
Range of Motion (ROM) of the Glenohumeral Joint [Mean (Standard Deviation); unit: degree] — 1. before intervention for all participants
  2. using a goniometer
  3. patient sitting on a stool with the arm at anatomical position
  4. worst: 0 degree
  5. best: 360 degree
  degree | 223.56 (42.111) | 203.05 (46.163) | 215.20 (44.555)

OUTCOME MEASURES:

1. Primary Outcome: Range of Motion (ROM) of the Glenohumeral Joint
Description: 1. before intervention for all participants
  2. using a goniometer
  3. patient sitting on a stool with the arm at anatomical position
  4. worst: 0 degree
  5. best: 360 degree
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | CPIHD | CRIHD
Number analyzed (Participants) | 32 | 22
degree | 261.95 (47.197) | 241.84 (57.304)

2. Secondary Outcome: Pain Measured by Visual Analogue Scale (VAS)
Description: 1. before intervention for all participants
  2. using 10cm horizontal visual analog scale
  3. best: 0cm (no pain)
  4. worst: 10cm (worst pain)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | CPIHD | CRIHD
Number analyzed (Participants) | 32 | 22
cm | 2.96 (2.89) | 5.03 (2.95)

ADVERSE EVENTS:
Arm/Group | CPIHD | CRIHD
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/22
Other Adverse Events (participants affected / at risk) | 0/32 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes